CLINICAL TRIAL: NCT03949244
Title: Effect of Nailfold Application of Latanoprostene Bunod on Nailfold Capillary Blood Flow
Brief Title: Nailfold Capillary Blood Flow With Latanoprost Bunod
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James Tsai, Professor and System Chair of Ophthalmology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GCO 18-2686
Record Dates: First submitted 2019-05-12; First posted 2019-05-14 (Actual); Results first posted 2021-08-23 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Glaucoma, Open-Angle
Keywords: Nailfold capillary imaging; Latanoprost bunod; Latanoprost
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Latanoprost; BOL 303259-X; Saline Solution; Microscopic Angioscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients will have baseline NFC blood flow measurements after application of cedar oil. Then the study team will use NF application of either normal saline, latanoprost 0.005% or LTB 0.024% in random sequence. The patient and imager will know which study article is applied. NFC blood flow will be remeasured after 15 minutes. Preliminary data on controls suggests that 15 minutes is sufficient time to see a change in blood flow. NF article application will occur on a specially designed well applied to the 4th digit of the non-dominant hand. Two masked observers will evaluate NFC blood flow.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Latanoprost 0.005% (Active Comparator): Latanoprost 0.005% drops to the nailfold.
  Interventions: Drug: Latanoprost 0.005%; Diagnostic Test: Nailfold capillaroscopy
- Latanoprost bunod 0.024% (Experimental): Latanoprost bunod 0.024% drops to the nailfold.
  Interventions: Drug: Latanoprost bunod 0.024%; Diagnostic Test: Nailfold capillaroscopy
- Normal saline 0.9% (Placebo Comparator): Normal saline 0.9% to the nailfold.
  Interventions: Drug: Normal saline 0.9%; Diagnostic Test: Nailfold capillaroscopy

INTERVENTIONS:
Drug: Latanoprost 0.005% — Latanoprost 0.005% will be applied to the nailfold and images of the blood flow in the nailfold capillaries will be acquired.
  Other Names: Xalatan
  Arms: Latanoprost 0.005%
Drug: Latanoprost bunod 0.024% — Latanoprost bunod 0.024% will be applied to the nailfold and images of the blood flow in the nailfold capillaries will be acquired.
  Other Names: Vyzulta; LTB
  Arms: Latanoprost bunod 0.024%
Drug: Normal saline 0.9% — Normal saline 0.9% will be applied to the nailfold and images of the blood flow in the nailfold capillaries will be acquired.
  Arms: Normal saline 0.9%
Diagnostic Test: Nailfold capillaroscopy — An imaging system and does not penetrate the skin. A video camera with a magnifying lens used for studying the movement of blood in small blood vessels at the nailfold of the 4th finger.
  Other Names: NFC

SUMMARY:
The purpose of this study is to look at the relationship of small blood vessels irregularities observed with an imaging system called video nailfold capillaroscopy in people with primary open-angle glaucoma. Nailfold capillaroscopy (NFC) is a video camera with a magnifying lens used for studying the movement of blood in small blood vessels. It is simple, safe and does not penetrate the skin. The skin fold that is at the tip of the finger is called the "nailfold". NFC has been used to assess blood vessel narrowing in patients with glaucoma.

DETAILED DESCRIPTION:
In this study, the study team investigates the effect of topically-applied latanoprostene bunod (LTB) on the blood flow at the nailfold of the 4th finger in patients with primary open angle glaucoma. LTB is a new anti-glaucoma eye drop which received FDA clearance in early November 2017. It has two components: the prostaglandin analog (PGA) which decreases intraocular pressure (IOP) by enhancing the drainage of the aqueous (the fluid in the front part of the eye) from the eye, and the nitric oxide (NO) moiety which naturally dilates arteries in the body. The capillaries at the nailfold are comparable to those of the optic nerve head, which makes them a reasonable surrogate for evaluation of the effect of LTB on the blood flow. Therefore, this study may provide indirect evidence for the beneficial effect of LTB on blood flow to optic nerve which can potentially save the optic nerve from glaucomatous damage. Primary open angle glaucoma is a progressive condition and is the most common cause of irreversible blindness worldwide. Primary open angle glaucoma (POAG) is a subset of the glaucomas defined by an open, normal appearing anterior chamber angle and raised intraocular pressure (IOP), with no other underlying disease.

In addition to LTB, the study team will use latanoprost (L), an-FDA approved PGA anti-glaucoma eye drop and normal saline (NS: the physiologic solution composed of 0.9% salt and water), as controls to make sure the effects of LPB on nail fold capillary blood flow is not due to its PGA (as L is) or due to the placebo effect (as NS is).

This study may also serve as background information for the development of new anti-glaucoma medications which can be injected into the eye to facilitate blood flow to the optic nerve.

ELIGIBILITY:
Inclusion Criteria:

* 40 years old to 80 years old
* All participants will have open angles and no signs of secondary glaucoma such as exfoliation syndrome
* Untreated intraocular pressure (IOP) may be ≤ 21mmHg or ≥ 21mmHg in both eyes
* The cup-to-disc ratio (CDR) ≥ 0.6 in both eyes and CDR asymmetry ≤ 0.2.
* POAG patients will have reliable Humphrey Visual Field (HVF) loss consistent with optic nerve damage
* POAG patients can have any stage of POAG and be on any form of treatment for their disease.
* Willingness to sign informed consent and comply with study procedures.

Exclusion Criteria:

* History of non-POAG forms of glaucoma
* Pregnancy
* Inability to give informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ritch, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- New York Eye and Ear Infirmary of Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Results of the study will be shared as publications in peer-reviewed journals and at scientific meetings. All data to be shared will be de-identified. Study subjects may request to learn the results of the study, which will be provided orally by the study staff, or they will be referred to any publications.
Time Frame: Results will be shared upon completion of the study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at New York Eye and Ear Infirmary of Mount Sinai
Groups:
- Latanoprost 0.005%: Latanoprost 0.005% drops applied to the nailfold and images of the blood flow in the nailfold capillaries acquired.
  Nailfold capillaroscopy: An imaging system and does not penetrate the skin. A video camera with a magnifying lens used for studying the movement of blood in small blood vessels at the nailfold of the 4th finger.
- Latanoprost Bunod 0.024%: Latanoprost bunod 0.024% drops applied to the nailfold and images of the blood flow in the nailfold capillaries acquired via nailfold capillaroscopy.
- Normal Saline 0.9%: Normal saline 0.9% to the nailfold and images of the blood flow in the nailfold capillaries acquired via nailfold capillaroscopy.
Period: Overall Study
Arm/Group | Latanoprost 0.005% | Latanoprost Bunod 0.024% | Normal Saline 0.9%
Started | 12 | 21 | 14
Completed | 12 | 21 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Latanoprost 0.005% | Latanoprost Bunod 0.024% | Normal Saline 0.9% | Total
Number analyzed (Participants) | 12 | 21 | 14 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.08 (5.95) | 66.95 (8.86) | 66.5 (8.50) | 66.84 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 8 | 29
  Male | 5 | 7 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 3 | 11
  Not Hispanic or Latino | 9 | 16 | 11 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 4 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 5
  White | 9 | 14 | 10 | 33
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: NFC Blood Flow at Baseline and 15 Minutes
Description: NFC blood flow at baseline and at 15 minutes after NF application to the 4th digit of the nondominant hand.
Time Frame: baseline and 15 minutes
Measure: Mean (Standard Deviation); unit: pL/s
Arm/Group | Latanoprost 0.005% | Latanoprost Bunod 0.024% | Normal Saline 0.9%
Number analyzed (Participants) | 12 | 21 | 14
pL/s
  Baseline | 72.52 (37.76) | 83.94 (78.31) | 93.01 (61.4)
  15 minutes | 60.50 (42.81) | 75.57 (44.68) | 69.70 (41.46)

ADVERSE EVENTS:
Time Frame: 15 minutes
Arm/Group | Latanoprost 0.005% | Latanoprost Bunod 0.024% | Normal Saline 0.9%
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/21 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/21 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/21 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT03949244/Prot_SAP_000.pdf